CLINICAL TRIAL: NCT01422642
Title: Do We Need High-Flexing Total Knee Arthroplasty to Improve the Survivorship and to Decrease the Incidence of Osteolysis? A Minimum of Ten Years of Follow-up
Brief Title: Do We Need High-Flexing Total Knee Arthroplasty to Improve the Survivorship and to Decrease the Incidence of Osteolysis?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPS-Flex vs LPS
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- legacy posterior stabilized high-flexion (Experimental): NexGen LPS-Flex total knee system
  Interventions: Device: legacy posterior stabilized high-flexion (NexGen LPS-Flex)
- legacy posterior stabilized standard (Experimental): standard NexGen LPS prosthesis
  Interventions: Device: legacy posterior stabilized standard (NexGen LPS)

INTERVENTIONS:
Device: legacy posterior stabilized high-flexion (NexGen LPS-Flex) — NexGen legacy posterior stabilized high-flexion (NexGen LPS-Flex) total knee system
  Other Names: NexGen LPS-Flex
  Arms: legacy posterior stabilized high-flexion
Device: legacy posterior stabilized standard (NexGen LPS) — NexGen legacy posterior stabilized standard (NexGen LPS) total knee system
  Other Names: NexGen LPS
  Arms: legacy posterior stabilized standard

SUMMARY:
The purpose of this study is to determine if there are any clinical or ROM differences in total knee arthroplasty with standard NexGen LPS prosthesis and NexGen LPS-Flex prosthesis.

DETAILED DESCRIPTION:
We therefore hypothesized: (1) the survival of the NexGen LPS-Flex prosthesis is better than standard NexGen LPS prosthesis; (2) knee function and range of motion after clinical assessment will be better in the NexGen LPS-Flex group; and (3) the incidence of osteolysis will be lower in the NexGen LPS-Flex prosthesis than standard NexGTne LPS prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 48 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2001-01; Primary Completion 2001-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | 10 years
  change in knee score will be compared with initial score, until mean follow up of 10.3 year

SECONDARY OUTCOMES:
Improvement in the range of motion | 10 years
  change in the range of motion of knee joint will be compared with the initial value, until mean follow up of 10.3 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University School of Medicine
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea